CLINICAL TRIAL: NCT06524154
Title: Effect of Verbal Positive Reinforcement, Contingent Escape and Rewarding on Behaviour of Children Undergoing Primary Molar Pulpotomy: a Randomized Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Khalid Aldhafeeri, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A01012023PP
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; Contingent Escape; Positive Reinforcement,; Pulpotomy; Behavior management

STUDY DESIGN:
Intervention Model Description: The study sample will comprise three groups, 14 children each randomly chosen. Group I: positive reinforcement, with praising the child with encouraging words and pleasing smiles.
  Group II: contingent escape, by giving some rest of the procedure while the child on the chair.
  Group III: rewarding the child with simple gifts like stickers at the end of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- positive reinforcement (Experimental): apply normal treatment with praising the child with encouraging words and pleasing smiles.
  Interventions: Behavioral: positive reinforcement
- contingent escape (Experimental): apply normal treatment with giving some rest of the procedure while the child on the chair.
  Interventions: Behavioral: contingent escape
- rewarding the child (Experimental): apply normal treatment with giving simple gifts like stickers at the end of the procedure.
  8
  Interventions: Behavioral: rewarding

INTERVENTIONS:
Behavioral: positive reinforcement — normal treatment with with praising the child with encouraging words and pleasing smiles.
  Arms: positive reinforcement
Behavioral: rewarding — normal treatment with giving simple gifts like stickers at the end of the procedure.
  Arms: rewarding the child
Behavioral: contingent escape — normal treatment with giving some rest of the procedure while the child on the chair.
  Arms: contingent escape

SUMMARY:
The purpose of this study to evaluate the effect of verbal positive reinforcement, contingent escape and rewarding on behaviour of children undergoing primary molar pulpotomy.

DETAILED DESCRIPTION:
this study evaluated Effect of Verbal Positive Reinforcement, Contingent Escape and Rewarding on Behaviour of Children Undergoing Primary Molar Pulpotomy

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 4 to 6 years of both sexes.
2. Children with behavior rating score 2,3 or 4 of Frankl 's behavior rating scale.
3. Children with carious lesions indicated for pulpotomy.
4. Restorable primary molars.

Exclusion Criteria:

1. Children with special health care needs.
2. Children suffering from systemic diseases.
3. Unrestorable tooth.
4. Extremely uncooperative children.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
RMS Pictorial Scale (RMS-PS) | 12 weeks
  The pictorial Scale (RMS) compromise's a row of five faces ranging from very happy very unhappy. The children will be asked to choose the face they feel like about themselves at that moment. The scale will be scored by giving a value of one to the very happy face and five to the very unhappy face

SECONDARY OUTCOMES:
Frankl Behavior Rating Scale | 12 weeks
  classified child's behavior into four groups according to the child's attitude and cooperation or lack of cooperation during dental treatment

OTHER OUTCOMES:
Pulse oximeter | 12 weeks
  To measure heart rate

CONTACTS AND LOCATIONS:
Overall Officials: khalid m aldhafeeri, master, Principal Investigator — Researcher of Pediatric Dentistry Faculty of Dentistry Mansoura University; abeer Mostafa A, Prof, Study Director — Professor and Head of Pediatric Dentistry Department- Department of Pediatric Dentistry- Faculty of Dentistry- Mansoura University; Rizk A Elagamy, PhD, Study Director — lecturer Pediatric Dentistry Department- Department of Pediatric Dentistry- Faculty of Dentistry- Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No